CLINICAL TRIAL: NCT05346185
Title: Association of Preoperative Sarcopenia on Postoperative Outcomes After Lung Cancer Surgery: Prospective Observational Study
Brief Title: Lung Cancer Surgery in Sarcopenia Patients With Old Age
Acronym: LUCAS-PEN
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, In Kyu Park, Professor, Seoul National University Hospital
Other Study IDs: 800-20210011
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Sarcopenia; Lung Cancer
Keywords: sarcopenia; lung cancer; surgery; long-term survival; complication; pulmonary function; quality of life
MeSH Terms: conditions — Sarcopenia; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The presence of sarcopenia before lung resection surgery might be an important factor of short-term and long-term prognosis in lung cancer patients. Through this study, investigators plan to demonstrate evidence whether sarcopenia is a useful clinical biomarker for risk stratification in elderly patients undergoing lung cancer surgery.

DETAILED DESCRIPTION:
Sarcopenia is a syndrome characterized by a decrease in the amount and function of skeletal muscle, and is known to have a prevalence of about 6-10% in 65 years of age or older and about 20-25% in 70 years of age or older. Recently, many studies have been conducted on the clinical importance of sarcopenia, and it has been reported that sarcopenia is significantly associated with a decline in quality of life and physical activity in the elderly population, as well as harmful clinical outcomes in postoperative patients and poor long-term outcomes in various solid cancer patients. Due to the promising result of lung cancer screening trial, lung cancer has been included in national cancer screening in South Korea since last year. As a result, more people are being diagnosed with lung cancer early. Furthermore, the number of patients having surgical resection for lung cancer is steadily growing, and as life expectancy rises, even older patients are increasingly considering surgical treatment. It's critical to appropriately assess risk in older individuals before and after surgery, and sarcopenia is considered a significant fartor for major surgery. According to studies on the association between sarcopenia and the postoperative clinical outcome of lung cancer surgery, sarcopenia evaluated by computed tomography has demonstrated to be associated with a poor surgical outcome and long-term prognosis. However, according to two recognized guidelines for sarcopenia (European Working Group on Sarcopenia in Elder People, and Asian Working Group for Sarcopenia), sarcopenia is supposed to comprehensively evaluate muscle mass, muscle strength, and physical activity. Regarding muscle mass, it is recommended to measure through dual energy-ray absoptiometery or bioelectrial impedance analysis. However, so far, there are no studies that have conducted an accurate evaluation of sarcopenia in elderly lung cancer patients and analyzed the relationship between them and the clinical outcome after lung cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients planning to perform curative surgery for confirmed lung cancer and pulmonary nodules suspected for lung cancer
* Patients or legal representatives who could understand and write written consent prior to the initiation of the clinical trial and are able to comply with the requirements for the clinical trial

Exclusion Criteria:

* Patients with treatment history for lung cancer or other solid cancer within 5 years (except patients with adenocarcinoma in situ for lung cancer)
* Patients who need simultaneous surgery with lung caner surgery for other accompanying diseases
* Patients who are not eligible to participate in the study judged by the researcher

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients above the age of 70 who are planning to undergo curative surgery for proven lung cancer or pulmonary nodules suspected for lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years after the day of lung cancer surgery
  survival status during the follow-up after the lung cancer surgery

SECONDARY OUTCOMES:
recurrence free survival | up to 5 years after the day of lung cancer surgery
  any recurrence or death during the follow-up after the lung cancer surgery
non-cancer related mortality | up to 5 years after the day of lung cancer surgery
  any death not related to lung cancer during the follow-up after the lung cancer surgery
postoperative change of pulmonary function | at postoperative 1 year, 5 year
  pulmonary function during the follow-up after the lung cancer surgery
postoperative complication rate | from the day of lung cancer surgery to the discharge after lung cancer surgery (up to 6 months)
  complication after lung cancer surgery
operative mortality | from the day of lung cancer surgery to the discharge after lung cancer surgery (up to 6 months)
  mortality related to lung cancer surgery
length of stays | from the day of lung cancer surgery to the discharge after lung cancer surgery (up to 6 months)
  length of hospital stays after lung cancer surgery
quality of life questionnaire | before the surgery, at postoperative 1 year, and at postoperative 5 year
  Five-level European quality of life Five Dimension (0 - 1, higher score means better outcome)
quality of life questionnaire | before the surgery, at postoperative 1 year, and at postoperative 5 year
  European quality of life visual analogue score ( 0 - 100, higher score means a better outcome)
geriatric depression scale questionnaire | before the surgery, at postoperative 1 year, and at postoperative 5 year
  Korean version geriatric depression scale (0-15, higher number indicates normal mood)
cognitive function questionnaire | before the surgery, and at postoperative 5 year
  Korean version Montreal Cognitive Assessment

CONTACTS AND LOCATIONS:
Overall Officials: In Kyu Park, MD, PhD, Principal Investigator — Seoul National University Hospital, Department of Thoracic and Cardiovascular Surgery
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Woo HS, Na KJ, Yun T, Park JH, Na B, Park S, Lee HJ, Kang CH, Kim YT, Park IK. Impact of sarcopenia on early surgical outcomes in elderly patients following lung cancer surgery: a prospective cohort study. J Thorac Dis. 2025 Oct 31;17(10):7838-7852. doi: 10.21037/jtd-2025-1375. Epub 2025 Oct 29. PMID 41229782